CLINICAL TRIAL: NCT00039325
Title: A Phase I/II Trial Testing Mart-1 Genetic Immunization In Malignant Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage IV or Recurrent Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069373; UCLA-9707074; NCI-G02-2077
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A - first dose for phase 1 (Experimental): A*0201 positive subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^6. Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine
- Arm B - dose increase for phase 1 (Experimental): A*0201 positive subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^7. Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine
- Arm C - A*0201+/DR*04+ subjects - Phase II (Experimental): Subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^7. Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine
- Arm D - A*0201+/DR*04- - phase 2 (Experimental): Subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^7. Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine
- Arm E - A*0201-/DR*04+ - phase 2 (Experimental): Subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^7. Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.
  Interventions: Biological: dendritic cell-MART-1 peptide vaccine

INTERVENTIONS:
Biological: dendritic cell-MART-1 peptide vaccine — Subjects will receive MART-1 adenovirus-transduced dendritic cells (DC)at dose of 10^6 (for arm A) or 10^7 (for arms B-E). Subjects will receive a total of three biweekly vaccinations given intradermally. If significant clinical or immunological response (to be defined later) is noted, subjects will be eligible for up to 6 additional monthly vaccine administrations.

SUMMARY:
RATIONALE: Vaccines made by inserting a laboratory-treated gene into a person's white blood cells may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of vaccine therapy and to see how well it works in treating patients with stage IV or recurrent malignant melanoma.

ELIGIBILITY:
Inclusion Criteria

* This study is confined to adults over the age of 18 with histologically proven malignant melanoma.
* MART-1, as assessed by either RT-PCR or by immunohistochemistry.
* Subjects must be typed for HLA-A*0201 for the phase I part of the study, and HLA-A*0201 and/or DR*04 for the phase II part.
* Stage with unresectable measurable melanoma (stage IV or stage III unresectable). Patients previously treated with any form of therapy (including chemotherapy, radiation therapy, immunotherapy or surgery) for either metastatic, relapsed or primary melanoma are eligible for this trial, provided that previous the previous treatment was completed > 30 days prior to first vaccine.
* Both male and female patients may be enrolled. Premenopausal females must have a negative pregnancy test prior to treatment.
* Karnofsky Performance Status greater than or equal to 70 percent, or ECOG greater than 2.
* No previous evidence of class 3 or greater New York Heart Association cardiac insufficiency or coronary artery disease.
* No previous evidence of opportunistic infection.
* A minimum of 30 days must have elapsed since the completion of prior chemotherapy, immunotherapy or radiation therapy.
* Adequate baseline hematological function as assessed by the following laboratory values within 30 days prior to study entry:

  * Hemoglobin > 9.0 g/dl.
  * Platelets > 100,000/mm3.
  * WBC > 3,000/mm3.
  * Absolute Neutrophil Count (ANC) > 1,000/mm3.
* Ability to give informed consent.

Exclusion Criteria

Patients who meet any one of the following criteria will be excluded from study entry:

* Lactating females: Females of child-bearing potential (pre-menopausal) must have a negative serum beta-HCG pregnancy test (within Day -7 to Day 0).
* Acute infection: any acute viral, bacterial, or fungal infection which requires specific therapy. Acute therapy must have been completed within 14 days prior to study treatment.
* HIV-infected patients, due to concerns in the ability to stimulate an effective immune response.
* Acute medical problems such as ischemic heart or lung disease that may be considered an unacceptable anesthetic or operative risk.
* Patients with any underlying conditions which would contraindicate therapy with study treatment (or allergies to reagents ).
* Patients with organ allografts.
* Uncontrolled CNS metastasis. Patients with CNS metastasis will be eligible if they have received CNS irradiation to control local tumor growth.
* Previous clinical evidence of an autoimmune disease.
* Concomitant Medication and Treatment

All allowed medications or treatments should be kept to a minimum and recorded. All questions regarding concomitant medications should be referred to the study chair or investigator.

Medications and Treatments Not Allowed

* Corticosteroids
* Chemotherapy
* Cyclosporin A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-03; Primary Completion 2005-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Optimal dose | 7 months

SECONDARY OUTCOMES:
Safety of administering MART-1 adenovirus transduced dendritic cells | 7 months
Immunological response (peptide-specific T cell generation, skin test immunohistology) | 7 months
Clinical response (disease improvement or disease progression) | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: James S. Economou, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States